CLINICAL TRIAL: NCT06611007
Title: Evaluation of the Safety of LipiodolⓇ Embolization in Symptomatic Digital Osteoarthritis Refractory to Conventional Treatment: a Pilot Study of 15 Patients
Brief Title: Evaluation of the Safety of LipiodolⓇ Embolization in Symptomatic Digital Osteoarthritis Refractory to Conventional Treatment
Acronym: EMBARDI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC23.0227; 2024-513361-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis
Keywords: Therapeutic embolization; Safety; Hand osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arterial embolization of the hand with Lipiodol (Experimental): The radial artery will be embolized with Lipiodol emulsified 3:1 with iodinated contrast medium (Optiray 300 mg/ml). The most painful hand according to VAS pain will be treated.
  Interventions: Drug: embolization therapy

INTERVENTIONS:
Drug: embolization therapy — Hand arterial embolization with Lipiodol in emulsion with iodinated contrast agent

SUMMARY:
The goal of this clinical trial is to evaluate the safety of arterial embolization using Lipiodol® in patients with symptomatic hand osteoarthritis refractory to conventional treatment. It will also learn about the efficacy of arterial embolization with Lipiodol® in reducing pain and improving hand function.

The main questions it aims to answer are:

* What are the side effects and complications associated with the Lipiodol® arterial embolization procedure?
* Does arterial embolization reduce pain intensity and improve hand function?

Researchers will evaluate patients over a 6-month period to assess the safety of Lipiodol® embolization and its impact on joint pain, swelling, and functional capacity. Participants will:

* Undergo arterial embolization with Lipiodol®
* Participate in regular follow-ups to monitor pain relief, hand function, and any side effects
* Have imaging studies to assess changes in joint vascularisation and damage

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years.
* Osteoarthritis of the hand according to American College of Rheumatology criteria 1990
* Osteoarthritis affecting at least two proximal and/or distal interphalangeal joints with a radiological Kellgren-Lawrence stage ≥ 2.
* Symptomatic osteoarthritis within the last 3 months.
* Visual analogue pain scale of the hand to be treated ≥ 40/100 mm (most painful hand).
* Inadequate response, adverse effects and/or contraindication to NSAIDs and non-opioid analgesics.
* Patient affiliated to french social security or a similar health assurance.

Exclusion Criteria:

* History of allergy to iodinated contrast media, LipiodolⓇ or poppies.
* Vasomotor disorders (Raynaud's syndrome, scleroderma, acrocyanosis).
* Stenosis (>50%) or known atheromatous arterial occlusion of the upper limbs.
* Obliterative arterial disease of the lower limbs at the critical ischaemia stage.
* Severe to end-stage chronic renal insufficiency (glomerular filtration rate < 30ml/min/1.73m2), dialysis or renal transplant.
* Arteritis such as thromboangiitis obliterans disease or other diseases
* Previous thrombosis/dissection of the radial artery.
* Chronic inflammatory rheumatic disease (rheumatoid arthritis, psoriatic arthritis, microcrystalline arthritis, etc.).
* Known hyperthyroidism or large multinodular goiter.
* Traumatic lesions, haemorrhages or chronic bleeding in the hand (not completely resolved within 3 months of the start of the lesion) requiring embolisation.
* Pregnant or breast-feeding.
* Patients covered by articles L1121-5 to L1121-8 of the French Public Health Code and/or who do not speak French.
* Patients in a period of exclusion or in the course of another interventional clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Number and Frequency of Embolisation-Related Adverse Events as Assessed by CTCAE | From embolization to 6 months after embolization
  The primary endpoint is the number and frequency of embolisation-related adverse events throughout the study period (6 months). Each adverse event will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) from grade 1 (mild) to grade 5 (fatal).

SECONDARY OUTCOMES:
Change Percentage of Participants Achieving at least a 50% improvement of pain Analog Visual Scale score at month 1 | baseline and month 1
  Percentage of patients with at least a 50% improvement in pain on the pain Analog Visual Scale score (0-100) of the treated hand compared to baseline, at month 1. VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The VAS is rated from 0 to 100 (no pain to extremely severe pain).
Change Percentage of Participants Achieving at least a 50% improvement of pain Analog Visual Scale score at month 3 | Baseline and Month 3
  Percentage of patients with at least a 50% improvement in pain on the pain Analog Visual Scale score (0-100) of the treated hand compared to baseline, at month 3. VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The VAS is rated from 0 to 100 (no pain to extremely severe pain).
Change Percentage of Participants Achieving at least a 50% improvement of pain Analog Visual Scale score at month 6 | Baseline and Month 6
  Percentage of patients with at least a 50% improvement in pain on the pain Analog Visual Scale score (0-100) of the treated hand compared to baseline, at month 1. VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patients marks. The VAS is rated from 0 to 100 (no pain to extremely severe pain).
Change From Baseline in Swollen Joints Counts at Month 1 | Baseline and Month 1
  Swollen joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Swollen Joints Counts at Month 3 | Baseline and Month 3
  Swollen joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Swollen Joints Counts at Month 6 | Baseline and Month 6
  Swollen joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Tender Joints Counts at Month 1 | Baseline and Month 1
  Tender joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Tender Joints Counts at Month 3 | Baseline and Month 3
  Tender joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Tender Joints Counts at Month 6 | Baseline and Month 6
  Tender joints of hand are indentified by clinical examination. Following joints are assessed : wrists, trapeziometacarpal joints, first to five metacarpophalangeal joints, first to five proximal interphalangeal joints, second to five distal interphalangeal joints
Change From Baseline in Cochin Hand Function Index score at Month 1 | From Baseline and Month 1
  Cochin Hand Function Index Score is a functional disability scale for hand comprising 18 questions on daily activities. This question is completed by the patient. Final score is obtained by adding the score of each question rated on a Likert scale from 0 (done without difficulty) to 5 (impossible to do).
Change From Baseline in Cochin Hand Function Index score at Month 3 | From Baseline and Month 3
  Cochin Hand Function Index Score is a functional disability scale for hand comprising 18 questions on daily activities. This question is completed by the patient. Final score is obtained by adding the score of each question rated on a Likert scale from 0 (done without difficulty) to 5 (impossible to do).
Change From Baseline in Cochin Hand Function Index score at Month 6 | From Baseline and Month 6
  Cochin Hand Function Index Score is a functional disability scale for hand comprising 18 questions on daily activities. This question is completed by the patient. Final score is obtained by adding the score of each question rated on a Likert scale from 0 (done without difficulty) to 5 (impossible to do).
Change From Baseline in Functional Index for Hand Osteoarthritis at Month 1 | From Baseline and Month 1
  The Functional Index for Hand Osteoarthritis (FIHOA) assesses hand osteoarthrits-related functional impairment scoring from 0 (no functional impairment) to 30 points (maximal impairment).
Change From Baseline in Functional Index for Hand Osteoarthritis at Month 3 | From Baseline and Month 3
  The Functional Index for Hand Osteoarthritis (FIHOA) assesses hand osteoarthrits-related functional impairment scoring from 0 (no functional impairment) to 30 points (maximal impairment).
Change From Baseline in Functional Index for Hand Osteoarthritis at Month 6 | From Baseline and Month 6
  The Functional Index for Hand Osteoarthritis (FIHOA) assesses hand osteoarthrits-related functional impairment scoring from 0 (no functional impairment) to 30 points (maximal impairment).
Change From Baseline in quick Disabilities of the Arm, Shoulder, and Hand at Month 1 | From Baseline and Month 1
  The QuickDASH (Disabilities of the Arm, Shoulder, and Hand) is a shortened version of the DASH questionnaire, designed to evaluate upper limb function and symptoms. It consists of 11 questions that measure physical function and symptoms related to daily activities, work, and leisure. Each item is scored on a 5-point scale, with higher scores indicating greater disability. The final score is calculated in accordance with the following formula: =((sum of n responses/n)-1)x25, where n represents the number of completed responses.
Change From Baseline in quick Disabilities of the Arm, Shoulder, and Hand at Month 3 | From Baseline and Month 3
  The QuickDASH (Disabilities of the Arm, Shoulder, and Hand) is a shortened version of the DASH questionnaire, designed to evaluate upper limb function and symptoms. It consists of 11 questions that measure physical function and symptoms related to daily activities, work, and leisure. Each item is scored on a 5-point scale, with higher scores indicating greater disability. The final score is calculated in accordance with the following formula: =((sum of n responses/n)-1)x25, where n represents the number of completed responses.
Change From Baseline in quick Disabilities of the Arm, Shoulder, and Hand at Month 6 | From Baseline and Month 6
  The QuickDASH (Disabilities of the Arm, Shoulder, and Hand) is a shortened version of the DASH questionnaire, designed to evaluate upper limb function and symptoms. It consists of 11 questions that measure physical function and symptoms related to daily activities, work, and leisure. Each item is scored on a 5-point scale, with higher scores indicating greater disability. The final score is calculated in accordance with the following formula: =((sum of n responses/n)-1)x25, where n represents the number of completed responses.
Change from Baseline in Hand grip strength at Month 1 | Baseline and Month 1
  Grip strength of the hand is assessed using a Grip Strength Hand Dynamometer. The result is expressed in kilograms.
Change from Baseline in Hand grip strength at Month 3 | Baseline and Month 3
  Grip strength of the hand is assessed using a Grip Strength Hand Dynamometer. The result is expressed in kilograms.
Change from Baseline in Hand grip strength at Month 6 | Baseline and Month 6
  Grip strength of the hand is assessed using a Grip Strength Hand Dynamometer. The result is expressed in kilograms.
Change from Baseline of Number and Severity of joint vascularization assessed by doppler Ultrasound at Month 1 | Baseline and Month 1
  Doppler vascularisation was assessed using a semi-quantitative score (0-3, 0: no vascularisation, 3: high vascularisation) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of joint vascularization assessed by doppler Ultrasound at Month 3 | Baseline and Month 3
  Doppler vascularisation was assessed using a semi-quantitative score (0-3, 0: no vascularisation, 3: high vascularisation) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of joint vascularization assessed by doppler Ultrasound at Month 6 | Baseline and Month 6
  Doppler vascularisation was assessed using a semi-quantitative score (0-3, 0: no vascularisation, 3: high vascularisation) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of synovitis assessed by Ultrasound at Month 1 | Baseline and Month 1
  Synovitis was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no synovitis, 3: significant synovitis) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of synovitis assessed by Ultrasound at Month 3 | Baseline and Month 3
  Synovitis was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no synovitis, 3: significant synovitis) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of synovitis assessed by Ultrasound at Month 6 | Baseline and Month 6
  Synovitis was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no synovitis, 3: significant synovitis) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of joint effusion assessed by Ultrasound at Month 1 | Baseline and Month 1
  Joint effusion was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no joint effusion, 3: high joint effusion) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of joint effusion assessed by Ultrasound at Month 3 | Baseline and Month 3
  Joint effusion was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no joint effusion, 3: high joint effusion) in acccordance with OMERACT guidelines.
Change from Baseline of Number and Severity of joint effusion assessed by Ultrasound at Month 6 | Baseline and Month 6
  Joint effusion was assessed using B-mode ultrasound and a semi-quantitative score (0-3, 0: no joint effusion, 3: high joint effusion) in acccordance with OMERACT guidelines.
Change from 6 months prior to inclusion in use of pain medication over the 6 months of study | From 6 months before inclusion to Month 6
  Pain medication will be described using analgesic level.
Change in the intensity of neovascularisation in the hand joints, as assessed by arteriography, from before embolisation to immediately after embolisation | Before and Immediately after embolisation
  A semi-quantitative assessment of neovascularisation (weak/moderate/important) before and after embolisation of the treated hand by analysing vascuralisation throw angiography is performed The following joints are evaluated : Trapezium-metacarpal joint, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, distal interphalangeal (DIP) joints 2-5.
Change From Baseline in Ghent University Scoring System (GUSS) at Month 6 | Baseline and Month 6
  The Ghent University Scoring System (GUSS) is a radiographic scoring method specifically developed to evaluate joint damage in hand osteoarthritis. It focuses on assessing both structural damage and remodeling features visible on hand X-rays. Erosive progression and signs of repair or remodelling are scored by indicating the proportion of normal subchondral bone, subchondral plate and joint space on an 11-point rating scale (range 0-100 with 10 unit increases). A lower score indicates greater damage or remodeling. The total score is the sum of these 3 scores for the joint under consideration.
Change in hand cutaneous microcirculation assessed by Laser Speckle Contrast Imaging (LSCI) before and during two hours post embolization | Before embolisation and 0, 15, 30, 45, 60, 75, 90, 105 and 120 minutes post embolisation
  A PeriCam PSI device (Perimed, Sweden) will be used to assess skin perfusion in both hands. The image size will be set at 30 x 20 centimetres and the acquisition speed at one image per second. The wavelength chosen will be 785 nm and the laser head will be positioned between 15 and 20 centimetres above the hands (with a resolution of ~ 6.9 pixels/ cm2). Cutaneous blood flow in the areas of interest will be expressed as PU (perfusion unit) and/or CVC (cutaneous vascular conductance). The area of interest will be the whole hand and the area around each hand joint.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Romand, MD, PhD, Principal Investigator — CHU Grenoble Alpes, site Sud, France
Locations (1):
- CHU Grenoble Alpes - Sud site, Échirolles, France

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual data and other informations as study protocole, informed consent form, clinical study report.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers to the corresponding author. The data will be shared on reasonable request after will be provided following review and approval of a research proposal and statistical analysis plan. A contract will be drawn up and signed to ensure, in particular, compliance with the RGPD rules, confidentiality.